CLINICAL TRIAL: NCT03769311
Title: A Window of Opportunity Trial of Cetuximab in Patients With Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Cetuximab in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW18098; P50DE026787 (NIH); NCI-2018-02990 (Other: NCI Trial ID); 2018-1232 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); Protocol Version 6/26/2020 (Other: UW Madison)
Record Dates: First submitted 2018-11-28; First posted 2018-12-07 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Single site, open label, window of opportunity study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pre-Operative Cetuximab Therapy (Experimental): Two weekly doses of pre-operative cetuximab during the interval between diagnostic HNSCC biopsy and surgery (~14 days), ensuring that no delay in standard of care (SOC) will occur. For dose #1, participants will receive cetuximab 400 mg/m2 via intravenous infusion over 2 hours (maximum infusion rate 10 mg/min) as per the standard of care loading regimen for cetuximab monotherapy. For dose #2, participants will receive cetuximab 250 mg/m2 via intravenous infusion over 1 hour (maximum infusion rate 10 mg/min) as per the standard of care dosing regimen for cetuximab monotherapy.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Monoclonal antibody against epidermal growth factor receptor (EGFR)
  Other Names: CTX; Erbitux

SUMMARY:
This clinical trial is for participants with head and neck squamous cell carcinoma who are scheduled to have their tumor surgically removed. The study involves obtaining baseline tissue from a clinical biopsy or research biopsy and measurement of circulating tumor cells before surgery to determine whether AXL protein expression pre-treatment correlates to clinical outcomes (change in tumor size) after two doses of cetuximab. The importance of this study is to describe if AXL expression can be used as a biomarker to predict clinical response to cetuximab (CTX) treatment.

DETAILED DESCRIPTION:
This is a window of opportunity trial evaluating the hypothesis that AXL levels correlate with clinical response to cetuximab in head and neck patients. Patients with head and neck squamous cell carcinoma who are scheduled to undergo surgical resection of their tumor and are candidates for cetuximab chemotherapy are eligible to participate.

Primary:

1. To test the hypothesis that low AXL correlates with clinical response to cetuximab in head and neck cancer patients

Secondary:

1. To further describe the safety of pre-operative administration of cetuximab

Correlative:

1. To correlate AXL expression with change in Ki67 following cetuximab in Head and Neck Cancer (HNC) patients
2. To examine other putative markers of cetuximab sensitivity such as HER3 and change in circulating tumor cells
3. To establish the first panel of patient-derived xenografts from patients with known sensitivity or resistance to cetuximab

Following informed consent, tumor tissue from the research biopsy and a blood draw for circulating tumor cells will be obtained. The participant will then receive two weekly doses of pre-operative cetuximab during the interval between diagnostic biopsy and surgery (~14 days), ensuring that no delay in standard of care (SOC) will occur.

For dose #1, participants will receive cetuximab 400 mg/m2 via intravenous infusion over 2 hours (maximum infusion rate 10 mg/min) as per the standard of care loading regimen for cetuximab monotherapy.

For dose #2, participants will receive cetuximab 250 mg/m2 via intravenous infusion over 1 hour (maximum infusion rate 10 mg/min) as per the standard of care dosing regimen for cetuximab monotherapy.

At the time of surgery, another blood draw will be obtained for analysis of circulating tumor cells, and a portion of the resected tumor will be obtained for study analysis.

Correlative studies will include the measurement of proteins hypothesized to be involved in cetuximab resistance such as AXL, Ki67, EGFR, and HER3 expression from both the biopsy and the surgical specimen. Blood will be analyzed for correlative analysis of circulating tumor cells. Tissue from the research biopsy will be utilized for participant-derived xenograft (PDX) development.

ELIGIBILITY:
Inclusion Criteria:

Informed consent: participants must be informed of the investigational nature of the study and must be able to sign a written informed consent.

* Inclusion criteria for research biopsy (screen)

  * Participants must have suspected or known clinical presentation of head and neck squamous cell carcinoma or a recurrence of head and neck squamous cell carcinoma after initial therapy. For newly suspected head and neck cancer, the procedure will obtain tissue for both standard of care biopsy and additional tissue for research.
  * Participants must have sufficient tumor volume (approximately 10 cc) to accommodate at minimum 2-3 core samples for the research biopsy. This will be approximated based on clinical evidence, such as physician visualization or palpitation.
  * Participants are required to consent to the TSB Biobank protocol (2016-0934) as part of this study.
  * Surgical management must be the chosen modality for management of the head and neck squamous cell cancer.

    * Other therapeutic modalities may follow, but surgery must be the choice for first therapy rendered.
* Inclusion criteria for cetuximab treatment:

  * Participants must have a biopsy proven, squamous cell carcinoma of the head and neck, excluding advanced cutaneous head and neck squamous cell carcinoma.
  * ECOG performance status £ 1
  * Women of childbearing potential (WOCP) must not be pregnant (confirmed by a negative urine/serum pregnancy test within 7 days of cetuximab treatment). In addition, a medically acceptable method of birth control must be used such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence during the study participation and for 6 months after last dose of study drug. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
  * Men who are not surgically or medically sterile must agree to use an acceptable method of contraception. Male participants with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant must agree to use condoms during the study and for 6 months post study drug. Total abstinence for the same study period is an acceptable alternative.
  * Participants with other concomitant malignancies are allowed to participate on the clinical trial as long as the surgical resection of the head and neck squamous cell carcinoma is clinically indicated.
  * Participants with metastatic disease are allowed to participate on the clinical as long as the surgical resection of the head and neck squamous cell carcinoma is clinically indicated.

Exclusion Criteria:

* Diagnosis of nasopharyngeal carcinoma, advanced cutaneous squamous cell carcinoma of the head & neck, and salivary gland tumors
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Prior chemotherapy, radiotherapy, or major surgery within 8 weeks of study enrollment or those who have not recovered (to grade ≤ 1 or baseline) from clinically significant adverse events due to agents administered more than 8 weeks earlier (alopecia and fatigue excluded). Clinical significance to be determined by the study investigator
* Prior cetuximab therapy is allowed so long as administered ³ 8 weeks ago.
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab
* Pregnancy, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment
* Ongoing or active infection, including active tuberculosis or known infection with the human immunodeficiency virus (HIV)
* Ongoing treatment with other investigational agents.
* Any of the following cardiac conditions:

  * uncontrolled or poorly-controlled arrhythmia or uncontrolled cardiac insufficiency uncontrolled or poorly-controlled hypertension (>180 mmHg systolic or > 130 mmHg diastolic)
* Any of the following conditions:

  * serious or non-healing wound, ulcer, or bone fracture
  * history of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 28 days of study enrollment
  * history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study enrollment
  * history of myocardial infarction, ventricular arrhythmia, stable/unstable angina, symptomatic congestive heart failure, coronary/peripheral artery bypass graft or stenting or other significant cardiac disease within 6 months prior to study enrollment
  * history of arterial or venous thrombosis/thromboembolic event, including pulmonary embolism within 6 months of study enrollment
  * any condition requiring the use of immunosuppression, excluding rheumatologic conditions treated with stable doses of corticosteroids
  * Use of herbal supplements (St. John's Wort, gingko biloba, etc.) within one week of cetuximab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bruce, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Wisconsin Carbone Cancer Center from April 2019 to March 2021.
Period: Overall Study
Arm/Group | Pre-Operative Cetuximab Therapy
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pre-Operative Cetuximab Therapy
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  20-29 | 1
  30-39 | 1
  40-49 | 2
  50-59 | 2
  60-69 | 6
  70-79 | 2
  80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Disease Site [Count of Participants; unit: Participants]
  Floor of Mouth | 3
  Tongue | 8
  Tonsil | 1
  Soft Palate | 1
  Other, unspecified parts of mouth | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Size
Description: The tumor size (via clinical measurements) will be measured from the time of diagnosis (pre-CTX) to after treatment with 2 doses of cetuximab and within 48 hours prior to surgery (post-CTX). Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Committee criteria will be used to define clinical response (partial response, progressive disease, or stable disease) prior to surgery.
Time Frame: up to 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Operative Cetuximab Therapy
Number analyzed (Participants) | 15
Participants
  Partial response | 1
  Progressive disease | 3
  Stable disease | 11

2. Primary Outcome: Objective Tumor Response Rate - AXL Expression
Description: The levels of AXL expression (low vs high, ranges from 0-4+ with 4+ meaning intense staining in the majority of cancer cells and 0 meaning no staining at all) at the time of diagnosis (pre-CTX) will measured and compared to change in the tumor size as reported in Primary Outcome Measure 1.
Time Frame: up to 42 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Pre-Operative Cetuximab Therapy
Number analyzed (Participants) | 14
score on a scale | 2.3 [1 to 4]

3. Secondary Outcome: Number of Hospital Re-admission for CTX-related Complications
Description: Hospital re-admission for wound healing, surgical complications, or infection that occur within 28 days after surgery will be categorized as definitely related, probably related, possibility related, unlikely related, or unrelated to cetuximab administration and will be reported as a number of participants.
Time Frame: within 28 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Operative Cetuximab Therapy
Number analyzed (Participants) | 15
Participants | 0

4. Other Pre Specified Outcome: Change in Ki67 From Pre- vs Post-CTX Treated Tumors
Description: Summary statistics of the change in Ki67 (ΔKi67), as established by the surgical specimen, will be reported for the response to cetuximab endpoint.
Time Frame: up to 30 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Correlation of Measures of Putative Markers of CTX Sensitivity
Description: Markers include: protein, RNA, circulating tumor cells with CTX response, measured by Ki67. Correlation between ΔKi67 and putative biomarkers will be analyzed as a continuous variable and will be tested using Pearson's correlation coefficient. Correlation between two biomarkers such as AXL and HER3 expression as continuous variables will be investigated using Pearson's correlation coefficient. Summary statistics will be used to report circulating tumor cells at each time point and the changes between time points. The association of change in circulating tumor cells with ΔKi67 (early response) will be explored graphically and with Pearson's correlation coefficient.
Time Frame: up to 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All AE's will be recorded from the time of informed consent until 28 days past last dose of study drug or day of surgery, whichever is first. SAE's will be recorded from the time of informed consent through 28 days past last dose of study drug or 28 days post-surgery, whichever is later. Up to 10 weeks on study.
Arm/Group | Pre-Operative Cetuximab Therapy
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Operative Cetuximab Therapy (N=15)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 4
Joint Aches (Musculoskeletal and connective tissue disorders) | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 1
Oral Pain (Gastrointestinal disorders) | 2
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03769311/Prot_SAP_000.pdf